CLINICAL TRIAL: NCT05626205
Title: PARO: Psycho-social Intervention With Paro Robotic Seal Focused on Patients With Dementia
Brief Title: Psycho-social Intervention With Paro Robotic Seal Focused on Patients With Dementia
Acronym: PARO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INRCA_006_2022
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease; Older Adults
Keywords: technology-based intervention; Alzheimer Disease; Dementia; Older Adults
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Experimental Group will receive for 12 weeks a robotic training with Paro robot combined with traditional training.
  Interventions: Device: PARO robot
- Control Group (No Intervention): The Control Group will receive only the traditional therapy.

INTERVENTIONS:
Device: PARO robot — PARO is an advanced interactive robot. It allows the documented benefits of animal therapy to be administered to patients in environments such as hospitals and extended care facilities where live animals present treatment or logistical difficulties. PARO has five kinds of sensors: tactile, light, audition, temperature, and posture sensors, with which it can perceive people and its environment. PARO can learn to behave in a way that the user prefers, and to respond to its new name.
  Arms: Experimental Group

SUMMARY:
The overall objective of the study is to evaluate the improvement in patient-perceived quality of life following the use of the Paro robot integrated with traditional intervention in the elderly with dementia.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the patient-perceived improvement in terms of quality of life through Quality of Life - Alzheimer's Disease (QoL-AD), following the use of the Paro robot, integrated with traditional intervention carried out within the IRCCS INRCA Alzheimer's Day Center.

The Secondary aims are the evaluation of the improvement in cognitive status of the elderly person with dementia, in terms of orientation, attentional-executive, mnestic and visuospatial functions, detected through the Addenbrooke's Cognitive Examination (ACE-R); the assessment of mood improvement in terms of reduction of anxiety and depression, detected through the Rating Anxiety In Dementia (RAID) scale and the Cornell Scale for Depression in Dementia (CSDD); the assessment of the elderly person's acceptance of the technology through Quebec User Evaluation of Satisfaction (QUEST 2.0), semi-structured interview and analysis of physiological activation during interaction, with the Noldus Face Reader system and direct observation by the operator; the analysis of behavioral symptomatology through Neuropsychiatric Inventory (NPI); the assessment of practitioner's acceptance of technology through Technology Acceptance Model (TAM) and the assessment of job quality through semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild-moderate dementia according to the Diagnostic and Statistical Manual of Mental Disorders (DSM V).
* MMSE between 10 and 24
* Attending the Alzheimer's Day Center since at least 3 months
* Presence of a caregiver

Exclusion Criteria:

* Severe sensory disabilities (visual and auditory)
* Comprehension difficulties
* History of syncopal episodes, epilepsy, and dizziness not controlled pharmacologically
* Severe autonomic system dysfunction
* Severe behavioral syndromes not compensated by medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-05 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
changes in quality of life | baseline, 12 and 24 weeks later
  This outcome will be assesed by the Quality of life in Alzheimer's Disease (QoL-AD) test. The QoL-AD is comprised of 13 items (physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole). Response options include 1(poor), 2(fair), 3(good) and 4 (excellent), for a total score of 13-52, with higher scores indicating better QoL.

SECONDARY OUTCOMES:
changes in cognitive status | baseline, 12 and 24 weeks later
  This outcome will be assessed by the Addenbrooke's Cognitive Examination (ACE-R). It contains5 sub-scores, each one representing one cognitivedomain: attention/orientation (18 points), memory(26 points), fluency (14 points), language (26 points)and visuospatial (16 points). ACE-R maximum score is 100, composed by the addition of the all domains. is scored out of 100, with a higher score denoting better cognitive function.
changes in mood | baseline, 12 and 24 weeks later
  This outcome will be assessed by the Rating Anxiety In Dementia (RAID). Rating should be based on symptoms and signs occurring during two weeks prior to the interview. No score should be given if symptoms result from physical disability or illness. Total score is the sum of items 1 to 18.
  A score of 11 or more suggests significant clinical anxiety.
changes in signs and symptoms of major depression | baseline, 12 and 24 weeks later
  This outcome will be assessed by the Cornell Scale for Depression in Dementia (CSDD). Information is elicited through two semi-structured interviews: an interview of an informant and an interview of the patient. Each item is rated for severity on a scale of 0-2 (0=absent, 1=mild or intermittent, 2=severe). The item scores are added. Scores above 10 indicate a probable major depression. Scores above 18 indicate a definite major depression. Scores below 6 as a rule are associated with absence of significant depressive symptoms.
changes in acceptance of the technology | baseline, 12 and 24 weeks later
  This outcome will be assessed by the technology through Quebec User Evaluation of Satisfaction (QUEST 2.0). The QUEST 2.0 evaluates the patient's satisfaction with various assistive technologies.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Bevilacqua, Principal Investigator — IRCCS INRCA
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

REFERENCES:
- [Derived] Bevilacqua R, Maranesi E, Felici E, Margaritini A, Amabili G, Barbarossa F, Bonfigli AR, Pelliccioni G, Paciaroni L. Social robotics to support older people with dementia: a study protocol with Paro seal robot in an Italian Alzheimer's day center. Front Public Health. 2023 Jun 21;11:1141460. doi: 10.3389/fpubh.2023.1141460. eCollection 2023. PMID 37415712